CLINICAL TRIAL: NCT00550251
Title: Does Acupressure Help Reduce Nausea and Vomiting in Palliative Care Patients? Formal Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sue Ryder Care (Other)
Responsible Party: Principal Investigator, Paul Perkins, Consultant in Palliative Medicine, Sue Ryder Care
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SRC2
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Nausea; Vomiting
Keywords: Nausea; Vomiting; Emesis; Palliative; Terminal; Cancer
MeSH Terms: conditions — Nausea; Vomiting; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupressure Bands (Active Comparator): Elasticated wrist bands with active bead pressing on Pericardium 6 acupressure points bilaterally.
  Interventions: Device: Acupressure Wrist Bands (Sea-Bands)
- Placebo (Placebo Comparator): Elasticated wrist bands without active bead.
  Interventions: Device: Placebo wristbands

INTERVENTIONS:
Device: Acupressure Wrist Bands (Sea-Bands) — Elasticated wrist bands with active bead pressing on Pericardium 6 acupressure points bilaterally.
  Other Names: Sea-Bands
  Arms: Acupressure Bands
Device: Placebo wristbands — Elasticated wrist bands without active bead.
  Other Names: Seaband Placebo
  Arms: Placebo

SUMMARY:
Pilot study completed - power calculation performed. Now formal double blind randomized study comparing active with placebo wristbands for nausea in palliative care patients to be carried out.

DETAILED DESCRIPTION:
Terminally ill hospice in-patients suffering with nausea will be randomized to active or placebo acupressure bands. The study will last 3 days and they will be allowed to continue regular or have PRN anti-emetics during the study.

Assessors and patients will both be blinded to whether they patients are receiving active or placebo bands.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of advanced cancer with an estimated prognosis of less than 1 year but more than 3 days.
2. Describe their nausea as at least moderate on a Likert scale OR at have had at least one vomit per day for the last three days.
3. Have an underlying cause for their nausea which is thought to be irreversible OR the patient has made an autonomous choice not to proceed with treatment for any potentially reversible cause (for example surgery for obstruction or drainage of ascites).
4. Can be male or female patients but must be over the age of 18.
5. Have signed a consent form prior to entering the study.
6. If patients are taking corticosteroids the dosage should be stable for 3 days before and during the trial.
7. Be thought to be well enough to complete the 3 day trial.

Exclusion criteria:

1. Arm lymphoedema.
2. Weakness, fatigue or confusion sufficient that patient is unable to take part.
3. Previous history of acupuncture/acupressure for nausea or vomiting, or history of use of acupressure by a close relative.
4. History of Parkinsonism or Parkinsonism on examination.
5. Patients will not be enrolled if they are sharing a room with another patient taking part in the study.
6. Patients who are unable to read or comprehend the questionnaire or Visual Analogue Scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2010-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Number of PRN Doses of anti-emetics needed | 3 days

SECONDARY OUTCOMES:
Visual Analogue Scale of nausea; duration of perceived nausea; number of vomits per 24 hours; volume of vomit per 24 hours; adverse effects of acupressure; measure of whether the patient felt the intervention helped. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Perkins, MB Bch MRCP, Study Director — Sue Ryder Care Leckhampton Court Hospice
Locations (1):
- Sue Ryder Care Leckhampton Court Hospice, Cheltenham, Gloucestershire, United Kingdom